CLINICAL TRIAL: NCT03967210
Title: Epidemiological, Clinical, Microbiological and Outcome Description of Patients With Klebsiella sp Meningitis
Acronym: KlebsieLCR
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: KlebsieLCR
Record Dates: First submitted 2019-05-24; First posted 2019-05-30 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Meningitis
MeSH Terms: conditions — Meningitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Klebsiella pneumoniae is implicated in the occurrence of severe pneumonia. Most Klebsiella pneumoniae infections are associated with care and occur in patients with compromised immune defenses. More recently, cases of hepatic abscess and acute community meningitis related to strains of Klebsiella pneumoniae have been reported. The mortality of these infections is important, most often due to a delayed diagnosis. The poor prognostic factors reported in the literature for very low numbers are: advanced age, coma, septic shock, glyceryachia <10mg / dL and proteinuria> 750 mg / dL. In addition, no study has specifically focused on the factors of occurrence and factors associated with Klebsiella sp. Indeed, meningitis related to Klebsiella pneumoniae seems to be a rare but probably underestimated event whose risk factors, clinical presentation, microbiological are little known and the treatment modalities of this severe infection are not codified.

ELIGIBILITY:
Inclusion Criteria:

* Man or Woman whose age ≥ 18 years
* Patient with meningitis Klebsiella sp., hospitalized in one of the hospitals of the Clinical Microbiology Group
* Francophone patient

Exclusion Criteria:

* Patient under tutorship or curatorship
* Patient deprived of liberty
* Patient under safeguard of justice
* Patient opposing his participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with meningitis Klebsiella sp., hospitalized in one of the hospitals of the Clinical Microbiology Group between 2008 and 2018.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2019-07-05 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-01-13 (Actual)

PRIMARY OUTCOMES:
Characterize meningitis with Klebsiella pneumoniae | Day 1
  This corresponds to characterize Klebsiella pneumoniae meningitis, portal entry, secondary infection, associated antibiotic and associated therapies and the clinical course of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Benoit PILMIS, MD, Study Director — Fondation Hôpital Saint-Joseph
Locations (18):
- France (18):
  - CHU Brest, Brest
  - CHU Caen, Caen
  - Hôpital henri Mondor, Créteil
  - CHU Lyon, Lyon
  - CHU Nantes, Nantes
  - CHU Nice, Nice
  - Hôpital Lariboisière, Paris
  - Groupe Hospitalier Paris Saint-Joseph, Paris
  - Hôpital Cochin, Paris
  - CHU Kremlin Bicetre, Paris
  - Hôpital Foch, Paris
  - Hôpital Necker Enfants Malades, Paris
  - Hôpital Sainte Anne, Paris
  - CHU Poitiers, Poitiers
  - CHU Reims, Reims
  - CHU Rennes, Rennes
  - CHU Strasbourg, Strasbourg
  - CHU Tours, Tours